CLINICAL TRIAL: NCT06954636
Title: Prognostic Potential of Olfactory Function in Glioblastoma: a Prospective Observational Study
Acronym: OLFGBM
Status: Recruiting | Type: Observational
Sponsor: Sied Kebir (Other)
Collaborators: Münster University Hospital, Germany (Unknown)
Responsible Party: Sponsor-Investigator, Sied Kebir, PD Dr. med., Head of Clinical Neuro-Oncology, University Hospital, Essen
Organization: University Hospital, Essen (Other)
Other Study IDs: 22-10501-BO
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma Multiforme, Adult; Glioblastoma or Gliosarcoma; Glioblastoma, Adult
Keywords: olfactory dysfunction; threshold test; identification test; glioblastoma; prognosis; observational study; olfactory function; neurocognition; quality of life
MeSH Terms: conditions — Glioblastoma; Gliosarcoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Newly-diagnosed glioblastoma cohort
  Interventions: Diagnostic Test: olfactory testing (threshold and identification test)
- Control cohort: Control group of patients with non-tumourous (neurological) diseases not primarily associated with an olfactory dysfunction
  Interventions: Diagnostic Test: olfactory testing (threshold and identification test)

INTERVENTIONS:
Diagnostic Test: olfactory testing (threshold and identification test) — In the identification test, 12 sniffin sticks are presented, which the patient has to name using a selection card with four terms each. Both nostrils are tested individually at each visit during the identification test. A correct answer scores one point. A maximum of 12 points is possible.
  The threshold test consists of 16 dilution levels. Each level contains one sniffin stick with odor and two blanks. All three sniffin sticks of a dilution level are presented to the patient one after the other with eyes closed. The patient must indicate which of the three sticks contains an odor. Depending on whether the patient gives the correct answer, the three sniffin sticks in the next higher or next lower level are presented next. A maximum of 16 points is possible.

SUMMARY:
The study aims to investigate the prognostic significance of olfactory function in patients with glioblastoma. We are examining olfactory function at various points during therapy and correlating the results with survival data. In addition, neurocognitive tests will be carried out to correlate the results of olfactory function with the patient's cognitive abilities. Investigations into the quality of life and psychological condition of the patients are also performed. In addition to the cohort of glioblastoma patients, there is a control cohort without tumor disease in which the olfactory testing is also carried out in order to have a comparison.

DETAILED DESCRIPTION:
Background: Olfactory impairment is frequent in glioblastoma and is associated with poor overall survival. However, earlier studies were limited by confounding of important predictive factors and the lack of long-term olfactory assessments to evaluate treatment-related neurotoxicity.

Aim: To determine whether olfactory function is an independent prognostic marker for survival, quality of life and neurocognitive outcome in glioblastoma.

Design: Prospective, multicenter cohort study with 64 glioblastoma patients and 64 comparable controls without tumor disease. Patients were stratified by baseline olfactory status, extent of resection, radiologic involvement of olfactory regions,O6-methylguanine DNA methyltransferase (MGMT) promoter methylation, age, and Karnofsky performance status.

Methods: Olfactory function will be serially assessed from diagnosis to treatment using Sniffin' Sticks (identification and threshold tests). Psychosocial assessments, neurocognitive testing and quality of life assessments will be performed at intervals. Coronal T2- and T1-weighted MRI scans will be evaluated independently by blinded neuroradiologists to identify olfactory involvement.

Next-generation sequencing will be used to investigate molecular correlates of hyposmia. As part of a parallel translational study, blood samples will be taken to analyze extracellular vesicles.

Olfactory testing:

In the identification test, 12 sniffin sticks are presented, which the patient has to name using a selection card with four terms each. Both nostrils are tested individually at each visit during the identification test. A correct answer scores one point. A maximum of 12 points is possible.

The threshold test consists of 16 dilution levels. Each level contains one sniffin stick with odor and two blanks. All three sniffin sticks of a dilution level are presented to the patient one after the other with eyes closed. The patient must indicate which of the three sticks contains an odor. Depending on whether the patient gives the correct answer, the three sniffin sticks in the next higher or next lower level are presented next. A maximum of 16 points is possible.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Newly-diagnosed glioblastoma (IDH wild-type)
* Never received prior chemotherapy
* Never received radiotherapy to the head or neck before
* KPS ≥ 70
* No history of severe head or brain trauma requiring ICU admission or classified as Glasgow Coma Scale grade 3
* No respiratory infection at the time of inclusion
* No significant aphasia

Exclusion Criteria:

* Presence of Neurodegenerative diseases (e.g. Parkinson's disease, Alzheimer's disease, Huntington's disease, Korsakoff's syndrome, Pick's disease, Shy-Drager syndrome)
* History of invasive tumors or surgery in the head or neck area, except for surgeries for non-invasive skin tumors (e.g. basal cell carcinomas)
* Permanent olfactory impairment following infections (e.g., influenza, coronavirus)
* Conditions that, in the examiner's judgment, could interfere with the participant's study compliance (e.g., schizophrenia)
* Language barriers likely to interfere with participation or comprehension of study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Newly-diagnosed glioblastoma
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From enrollment to 2 years after the end of radiotherapy
  Overall survival in relation to olfactory function

SECONDARY OUTCOMES:
Progression free survival | From enrollment to 2 years after the end of radiotherapy
  Progression free survival in relation to olfactory function
Neurocognition | From enrollment to 2 years after the end of radiotherapy
  Neurocognition in relation to olfactory function
  The following tests are used for neurocognition testing:
  * Immediate and delayed story recall from the Rivermead Behavioural Memory Test
  * Number span (forward and backward) and block span (forward and backward) from the Wechsler Memory Scale
  * Phonemic word fluency from the Regensburg Word Fluency Test (phonemic)
  * Trail Making Test A and B
Quality of Life (QoL) | From enrollment to 2 years after the end of radiotherapy
  Quality of Life in relation to olfactory function
  The following questionnaires are used to assess quality of life:
  * EORTC QLQ-C30 (Version 3.0; Part A with 28 questions on a Likert scale, 28 to 112 points, Higher score means lower quality of life; Part B with 2 questions on a Likert scale, 2 to 14 points, Lower score means lower quality of life )
  * EORTC QLQ-BN20 (20 questions on a Likert scale; 20 to 80 points; Higher score means lower quality of life)
Psychological condition | From enrollment to 2 years after the end of radiotherapy
  Psychological well-being in relation to olfactory function
  The following psychiatric questionnaires are used:
  * Patient Health Questionnaire-8 (PHQ-8):
    8 questions on a Likert scale, score 0 to 24, higher score indicate more depression
  * Generalized Anxiety Disorder 7 (GAD-7):
    7 questions on a Likert scale, score 0 to 21, higher score indicate more anxiety
  * National Comprehensive Cancer Network (NCCN) Distress Thermometer:
  Score 1 to 10, higher score indicate more distress

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Essen, Department of Neurology, Division of Clinical Neuro-Oncology, Essen
  - Department of Neurosurgery, Münster

IPD SHARING:
Plan to Share IPD: Yes
Clinical Data from the other study centers will be transferred pseudonymously to the study headquarters in Essen. Only pseudonymized data is also used for accompanying scientific projects.

REFERENCES:
- [Background] Hummel T, Sekinger B, Wolf SR, Pauli E, Kobal G. 'Sniffin' sticks': olfactory performance assessed by the combined testing of odor identification, odor discrimination and olfactory threshold. Chem Senses. 1997 Feb;22(1):39-52. doi: 10.1093/chemse/22.1.39. PMID 9056084
- [Background] Hummel T, Konnerth CG, Rosenheim K, Kobal G. Screening of olfactory function with a four-minute odor identification test: reliability, normative data, and investigations in patients with olfactory loss. Ann Otol Rhinol Laryngol. 2001 Oct;110(10):976-81. doi: 10.1177/000348940111001015. PMID 11642433
- [Background] Kebir S, Hattingen E, Niessen M, Rauschenbach L, Fimmers R, Hummel T, Schafer N, Lazaridis L, Kleinschnitz C, Herrlinger U, Scheffler B, Glas M. Olfactory function as an independent prognostic factor in glioblastoma. Neurology. 2020 Feb 4;94(5):e529-e537. doi: 10.1212/WNL.0000000000008744. Epub 2019 Dec 12. PMID 31831598
- [Background] Walker IM, Fullard ME, Morley JF, Duda JE. Olfaction as an early marker of Parkinson's disease and Alzheimer's disease. Handb Clin Neurol. 2021;182:317-329. doi: 10.1016/B978-0-12-819973-2.00030-7. PMID 34266602
- [Derived] Oster C, Matyar A, Schmidt T, Hummel T, Hattingen E, Jokisch M, Jokisch D, Grieger J, Cappello G, Kizina K, Lazaridis L, Ahmadipour Y, Rauschenbach L, Stuschke M, Pottgen C, Guberina N, Tertel T, Giebel B, Dreizner GL, Barbato F, Skoda EM, Scheffler B, Muther M, Herrmann K, Kleinschnitz C, Sure U, Deuschl C, Glas M, Kebir S. Decoding glioblastoma survival: unraveling the prognostic potential of olfactory function in a prospective observational study. Neurol Res Pract. 2025 Jul 24;7(1):51. doi: 10.1186/s42466-025-00410-2. PMID 40708059